CLINICAL TRIAL: NCT01728740
Title: Randomized, Non-blinded Crossover Study to Establish the Bioequivalence Between Fixed Dose Combination (FDC) and Loose Combination of Acarbose and Metformin and to Investigate the Potential for a Drug-drug Interaction Following Single Oral Dosing in Healthy Adult Male Subjects
Brief Title: Bioequivalence Study for Acarbose / Metformin FDC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head of Clinical Sciences, Bayer Healthcare AG
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 15420
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Bioequivalence; Acarbose; Metformin; FDC
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acarbose/Metformin FDC (Experimental): Day 0: oral sucrose load (75 g sucrose dissolved in 225 mL water) without Acarbose/Metformin FDC; Day 1: oral sucrose load plus single dose of 1 tablet Acarbose/Metformin FDC (containing 50 mg Acarbose and 500 mg Metformin)
  Interventions: Drug: Acarbose/Metformin FDC (BAY81-9783)
- Acarbose+Metformin (Active Comparator): Day 0: oral sucrose load (75 g sucrose dissolved in 225 mL water) without loose combination of Acarbose and Metformin; Day 1: oral sucrose load plus single dose of 1 tablet each of a loose combination of Acarbose 50 mg and Metformin 500 mg
  Interventions: Drug: Acarbose (Glucobay, BAYG5421); Drug: Metformin
- Acarbose (Active Comparator): Day 0: oral sucrose load (75 g sucrose dissolved in 225 mL water) without comedication; Day 1: oral sucrose load plus single dose of 1 tablet Acarbose 50 mg
  Interventions: Drug: Acarbose (Glucobay, BAYG5421)
- Metformin (Active Comparator): Day 0: oral sucrose load (75 g sucrose dissolved in 225 mL water) without comedication; Day 1: oral sucrose load plus single dose of 1 tablet Metformin 500 mg
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Acarbose/Metformin FDC (BAY81-9783) — Acarbose/Metformin FDC (BAY81-9783)50mg/500mg, oral, single dose
  Arms: Acarbose/Metformin FDC
Drug: Acarbose (Glucobay, BAYG5421) — Acarbose (Glucobay, BAYG5421) 50mg, oral, single dose
  Arms: Acarbose; Acarbose+Metformin
Drug: Metformin — Metformin 500mg, oral, single dose
  Arms: Acarbose+Metformin; Metformin

SUMMARY:
To establish the bioequivalence between Acarbose / Metformin FDC (50mg / 500mg) and loose combination of Acarbose (Glucobay) (50mg) and Metformin (Glucophage) (500mg).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI): 18 to 28 kg/m2 (inclusive)
* Results of Glycosylated Hemoglobin A1c (HbA1c) value are within the normal range (4.3-5.6%, inclusive)
* Results of the 75 g oral glucose tolerance test (OGTT) during screening show:

  * Blood glucose before OGTT <110 mg/dL.
  * Blood glucose 1 hour after glucose loading <180 mg/dL
  * Blood glucose 2 hours after glucose loading <140 mg/dL

Exclusion Criteria:

* A history of relevant diseases of internal organs (diabetes mellitus, Ileus, Ileus-like symptoms, diseases that may significantly jeopardize body systems
* Febrile illness within 1 week before drug administration
* Family history of diabetes (within the second degree of relationship)
* Known drug hypersensitivity or idiosyncrasy
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Habitual medication including Chinese herbal drugs
* Intake of any drugs within 2 weeks of drug administration of period 1
* Regular daily consumption of more than 1 L of usual beer or the equivalent quantity of approximately 40 g of alcohol in another form
* Donation of more than 150 mL of blood within 4 weeks before the screening examination
* Participation in another clinical trial within 4 weeks before the screening examination

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Ratio of postprandial maximum concentration (Cmax) of plasma glucose following sucrose load with (Day 1) and without acarbose (Day 0) | within 4 hours after sucrose load
Ratio of postprandial Area Under the Curve (AUC(0 4)) of plasma glucose following sucrose load with (Day 1) and without acarbose (Day 0) | within 4 hours after sucrose load
Cmax of metformin | within 24 hours after dosing
AUC(0-tn) of metformin | within 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Seoul, South Korea